CLINICAL TRIAL: NCT03564080
Title: An Investigation Into the Feasibility of Incorporating an Exercise Rehabilitation Programme for People With Peripheral Artery Disease Into an Already Established Cardiac Rehabilitation Service.
Brief Title: Assessing the Feasibility of Including Patients With Peripheral Artery Disease in to an Established Cardiac Rehabilitation Service.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salford (Other)
Collaborators: Northern Care Alliance NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Edward Caldow, Post Graduate Student, University of Salford
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSR1617-184
Record Dates: First submitted 2018-02-05; First posted 2018-06-20 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Peripheral Arterial Disease; Cardiovascular Diseases; Intermittent Claudication; Coronary Artery Disease
Keywords: exercise rehabilitation; supervised exercise programmes
MeSH Terms: conditions — Peripheral Arterial Disease; Cardiovascular Diseases; Intermittent Claudication; Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: Non-randomised control trial assessing feasibilty of new treatment method - combined supervised exercise programme
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control - PAD (No Intervention): This group of patients will complete the 'standard care' of supervised exercise as recommended by NICE.
- Combined - PAD and CAD (Experimental): This group of PAD patients will exercise alongside CAD patients in an established supervised exercise programme (Cardiac Rehabilitation).
  Interventions: Other: Combined - PAD and CAD

INTERVENTIONS:
Other: Combined - PAD and CAD — 12-week supervised exercise programme in a hospital setting
  Arms: Combined - PAD and CAD

SUMMARY:
This study will investigate if patients with peripheral artery disease (PAD) can be successfully incorporated into an already existing Cardiac Rehabilitation programme. One group of PAD patients will exercise as a group, and the other group will exercise alongside patients with coronary artery disease (CAD).

DETAILED DESCRIPTION:
Peripheral artery disease (PAD) is a progressive disease that occurs as the result of atherosclerotic plaque formation in the major arteries of the leg (Mays, Casserly and Regesteiner, 2013). The main presenting symptom of PAD is intermittent claudication (IC) - exertional pain or discomfort in the calf, thigh or buttock that is relieved with rest. The presence of PAD is a very powerful marker of cardiovascular risk and preventable cardiovascular deaths. Following the initial diagnosis of PAD, for those patients without coronary artery disease the risk of systemic morbidity or mortality in the next 5 years is 50% (AACVPR, 2013). In 2012, the National Institute for Health and Care Excellence (NICE) issued guidelines stating that supervised exercise programmes (SEPs) should be offered as first-line treatment for people diagnosed PAD. However, there is a national shortage of dedicated SEPs for PAD patients that UK vascular specialists can refer patients to. There has been suggestion that an already established network of Cardiac Rehabilitation (CR) departments within the United Kingdom (UK) could cater for this group of patients, as they already have facilities and staff in place. To date, there has been no investigation into whether this would be successful. This research project would investigate if CR programmes could get the same outcomes for PAD patients as a stand-alone PAD rehabilitation programme. The study would investigate the possible positive and negative impact on both the PAD and CR patient groups in attending a combined rehabilitation programme of exercise and education. It will also look at the perceptions of the participants regarding the treatment programme itself.

ELIGIBILITY:
Inclusion Criteria:

* General criteria As part of this study participants will be required to wear an accelerometer on the first week and last week of the 12 week study. The accelerometer will be kept in place by a medical dressing (e.g. Tegederm). People with an existing skin condition such as psoriasis or eczema that would be affected by the application of a medical dressing will be excluded from the study.

All participants must be able to start the incremental shuttle walk test (walking speed of 1.8kph, 1.1 mph).

All participants must be able to engage in the exercises prescribed in the programme

Inclusion Criteria - PAD patients:

All patients recruited will have had a recent diagnosis (0 - 12 months) of PAD made by either a vascular surgeon, vascular specialist nurse or specialist podiatrist.

Inclusion Criteria - CAD patients:

All patients recruited to the CR group will have had a recent diagnosis (0-12 months) of CAD (angina, myocardial infarction (MI), or coronary artery bypass graft (CABG) or valve surgery).

Exclusion Criteria:

* Exclusion criteria - PAD patients:

Any patient who has had previous intervention for PAD e.g. balloon angioplasty, stent, bypass or medication, or who have previously completed an SEP will be excluded from the study. This is due to the possibility of previous interventions having an impact on patient perceptions.

Participants who are on medication for PAD (e.g. naftidrofuryl oxalate) will also be excluded from the study as this can increase symptom management and improve functional capacity.

Any PAD patient who also has a diagnosis of other cardiovascular conditions such as CAD or stroke, or chronic heart failure will be excluded from this study, as the investigation is looking at the specific improvements in PAD, not CAD gains.

Exclusion criteria - CAD patients:

Any patient who has had previous diagnosis of PAD will be excluded from the study, as this may mask any gains in improvement due to CAD-specific rehabilitation in the CAD group (Tam et al., 2016).

Any participant who has unstable CAD (e.g. unstable angina) will be excluded from the study as this is a contraindication partaking in structured exercise programme (BACPR, 2012).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-07-18 (Actual); Primary Completion 2019-10-28 (Actual); Study Completion 2022-09-11 (Actual)

PRIMARY OUTCOMES:
Walking distance | 12 weeks
  Initial and maximal pain free walking distances are measured using a Incremental Shuttle Walk Test. The symptoms of claudication pain are identified using the American Association of Cardiovascular and Pulmonary Rehabilitation (AACVPR) 0-4 Claudication scale. 0 is no claudication; 1 is initial pain; 2 is moderate pain; 3 is severe; 4 is maximal pain.

SECONDARY OUTCOMES:
Walking Impairment Questionnaire | 12 weeks
  Patient's perceived walking distance and speed related to their claudication pain. Participants rate the distance and speed they are able to walk at. The distances are separated in to the amounts of blocks they can walk (with and without impairment). They then rate the speed they can walk 100 yards. The lower the score the worse the perceived limitation of their claudication symptoms.
King's College Vascular Quality of Life Questionnaire (VascQual) | 12 weeks
  Disease-specific quality of life questionnaire. The questionnaire is 25-item questionnaire subdivided into five domains: pain (4 items), symptoms (4 items), activities (8 items), social (2 items), and emotional (7 items). The higher the score the lower the health-related quality of life.
Free-living physical activity levels | 12 weeks
  Accelerometer data recording activity levels outside of rehabilitation programme
Hospital Anxiety and Depression Scale | 12 weeks
  The is a generic quality of life questions that assesses levels of anxiety and depression. There are 14 questions questions in total, 7 questions on anxiety and 7 on depression. Each question has an answer rating from 0-3, with 0 being no evidence of anxiety/depression, and 3 being maximum score. The total score for anxiety and depression are added (but anxiety and depression scores are not combined) to see the total reading for anxiety and depression. If 11 or above is scored in either anxiety or depression, then referral to appropriate health care professional is discussed with participant.

CONTACTS AND LOCATIONS:
Locations (1):
- Salford Royal NHS Foundation Trust, Salford, Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (3):
  • Study Protocol (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03564080/Prot_000.pdf
  • Statistical Analysis Plan (2017-08-16): https://cdn.clinicaltrials.gov/large-docs/80/NCT03564080/SAP_001.pdf
  • Informed Consent Form (2018-06-11): https://cdn.clinicaltrials.gov/large-docs/80/NCT03564080/ICF_002.pdf